CLINICAL TRIAL: NCT01175447
Title: A Phase I Study of S-1 With Concurrent Radiotherapy in Elderly Patients With Esophageal Cancer
Brief Title: S-1 and Radiotherapy in Elderly Patients With Esophageal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, JYongling, MD, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH07
Record Dates: First submitted 2010-07-31; First posted 2010-08-04 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Esophageal Cancer
Keywords: S-1; radiation; esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiotherapy with S-1 (Experimental): radiation 54Gy over 30 fractions,and concurrent with s-1 on days 1-14 and 29-42
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — S-1 was administered on days 1-14 and 29-42 at the following dosages: 60, 70, and 80mg/m(2)/day

SUMMARY:
Elderly patients with esophageal cancer will receive thoracic radiation therapy 54Gy over 30 fractions, and concurrent with s-1 on days 1-14 and 29-42 at the following dosages: 60, 70, and 80 mg/m(2)/day.

DETAILED DESCRIPTION:
Purpose:evaluated the dose-limiting toxicity and recommended dose of S-1 for a future phase II study when administered concurrently with thoracic radiation in elderly patients (>70 years old) with esophageal Cancer.

Methods:S-1 was administered on days 1-14 and 29-42 at the following dosages: 60, 70, and 80mg/m(2)/day. Thoracic radiation therapy was administered in 1.8Gy fractions five times weekly to a total dose of 54 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented diagnosis of esophageal Cancer
* Disease must be encompassed in a radiotherapy field.Patients with celiac, perigastric, mediastinal or supraclavicular adenopathy are eligible
* age:70-85 years
* Written informed consent.
* Performance status of 0 to 2
* Neutrophil count >1.5 x 10 to the 9th power/L and platelets > 100 x 10 to the 9th power/L.
* Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN) Alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN (or less than or equal to 5 times ULN in case of known liver involvement
* Renal: Serum Creatinine less than or equal to 1.5 times upper limit of normal (ULN)

Exclusion Criteria:

* Evidence of tracheoesophageal fistula, or invasion into the trachea or major bronchi.
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior systemic chemotherapy or radiation therapy for esophageal cancer

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of s-1 in combination with thoracic radiotherapy in elderly patients (> 70 years old) with esophageal Cancer | 3 months per patient
  the MTD will be defined as the maximum dose level at which no more than one subject out of six experiences a dose-limiting toxicity (DLT) during treatment.

SECONDARY OUTCOMES:
Objective response rate (e.g. complete response [CR], partial response [PR], stable disease [SD], or progressive disease [PD]). | dependent upon results

CONTACTS AND LOCATIONS:
Overall Officials: Xianghui Du, MD, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Ji Y, Qiu G, Sheng L, Sun X, Zheng Y, Chen M, Du X. A phase I dose escalation study of S-1 with concurrent radiotherapy in elderly patients with esophageal cancer. J Thorac Dis. 2016 Mar;8(3):451-8. doi: 10.21037/jtd.2016.02.70. PMID 27076940